CLINICAL TRIAL: NCT00310258
Title: Drug Abuse Prevention: A Mother-Daughter Intervention
Brief Title: Drug Use Prevention Among Girls Through a Mother-Daughter Intervention
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: girls & drugs; 5R01DA017721-02 (NIH)
Record Dates: First submitted 2006-03-30; First posted 2006-04-03 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2006-03

CONDITIONS: Adolescent Behavior
MeSH Terms: conditions — Adolescent Behavior

INTERVENTIONS:
Behavioral: Drug use prevention intervention

SUMMARY:
This study will develop and test drug use prevention strategies for low-income, minority girls. Gender-specific substance use rates, risk and protective factors, and health outcomes highlight the need for interventions aimed at girls. Girls and boys share a number of risk factors, yet some factors are more salient for one gender. Girls and boys may also be affected differently by the same risk factors. Intervention planned for this study emphasizes risk and protective factors that impact girls. Our intervention will build mother-daughter communication and closeness; enhance girls' self-efficacy and body esteem; nurture girls' conflict management, problem-solving, stress reduction, and refusal skills; correct perceived norms; build social supports; and establish patterns of parental monitoring and supervision. We hypothesise that girls who receive GSI will have lower 3-year follow-up rates of substance use than girls who receive no intervention.

The study will occur in three phases. In a 12-month preparation phase, we will refine and complete intervention and measurement protocols, recruit subjects and randomly assign girls and mothers to study arms, and pretest girls and mothers. A 12-month implementation phase will initiate field operations of the clinical trial, including intervention delivery, process data collection, and posttests. Follow-up in the last 36 months will involve longitudinal measurements of girls and mothers, booster session development and delivery, and data analyses.

DETAILED DESCRIPTION:
The study has two primary and seven secondary aims.

Primary Aims:

* 1. Develop a family-based girl-specific intervention (GSI) to prevent substance use.
* 2. Test the efficacy of GSI.

Secondary Aims:

* 3. Test GSI to improve mediating factors of girls' mother-daughter affective quality, coping, refusal skills, mood management, conflict resolution, problem solving, self-efficacy, body esteem, normative beliefs, social supports, and mother-daughter communication.
* 4. Examine the effects of mediating factors on girls' substance use behavior.
* 5. Test GSI to improve mothers' use of family rituals, rules against substance use, child management, mother-daughter affective quality, and communication with their daughters.
* 6. Examine the effects of mother' outcomes on their daughters' substance use behavior.
* 7. Test the effects of dose on participants' outcomes.
* 8. Determine if GSI has differential outcomes related to ethnic-racial group profile.

  9. Quantify the costs of intervention development and delivery.

ELIGIBILITY:
Inclusion Criteria:

* girls ages 11 to 13 years old at pretest and their mothers who have access to a private computer

Exclusion Criteria:

-

Ages: 11 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000
Dates: Start 2005-04; Study Completion 2006-02

PRIMARY OUTCOMES:
Scores on substance use behavior at posttest, and annually for 3 years after posttest.

SECONDARY OUTCOMES:
scores on mediating variables at posttest, and annually for 3 years after posttest.
closeness with mother
coping skills
refusal skills
depression (mood)
conflict resolution
problem solving
self-efficacy
body image
normative beliefs

CONTACTS AND LOCATIONS:
Overall Officials: Steven Schinke, Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University School of Social Work, New York, New York, United States

REFERENCES:
- [Result] Schinke S, Di Noia J, Schwinn T, Cole K. Drug abuse risk and protective factors among black urban adolescent girls: a group-randomized trial of computer-delivered mother-daughter intervention. Psychol Addict Behav. 2006 Dec;20(4):496-500. doi: 10.1037/0893-164X.20.4.496. PMID 17176186